CLINICAL TRIAL: NCT04006483
Title: A Review of Meta-Analyses on Bioavailable Stannous Fluoride Dentifrices: Effects on Dental Plaque
Brief Title: Meta-analysis of Stannous Fluoride and the Effects on Dental Plaque
Status: Completed | Type: Observational
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019SnF2PlaqueAnalysis
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stannous Fluoride Dentifrice: Twice daily brushing
  Interventions: Drug: Stannous fluoride dentifrice
- Positive control dentifrice: Twice daily brushing
  Interventions: Drug: Positive control dentifrice
- Negative control dentifrice: Twice daily brushing
  Interventions: Drug: Negative control dentifrice

INTERVENTIONS:
Drug: Stannous fluoride dentifrice — Stannous fluoride (0.454%) dentifrice
  Groups: Stannous Fluoride Dentifrice
Drug: Positive control dentifrice — Positive control dentifrice containing (0.3%) triclosan.
  Groups: Positive control dentifrice
Drug: Negative control dentifrice — Negative control dentifrice containing either sodium fluoride (0.243%) or sodium monofluorophosphate (0.76%)
  Groups: Negative control dentifrice

SUMMARY:
The aim of this 18 study analysis was to compare the effect of bioavailable stannous fluoride (SnF2) dentifrices when used up to 3 months on dental plaque relative to a positive or negative control dentifrice.

ELIGIBILITY:
Subjects were excluded from this study for the following reasons;

* pregnancy,
* rampant caries,
* severe periodontitis,
* at discretionary of the Principal Investigator.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This meta-analysis includes healthy adult male and females.
Sampling Method: Probability Sample
Enrollment: 2359 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Dental Plaque Scores | Up to 12 weeks
  Change from baseline as measured by mean plaque score reduction from baseline (via Quigley-Hein, Turesky Modification Index or Rustogi Modification of the Navy Plaque index).

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple P&G Investigation Clinical Sites, Cincinnati, Ohio, United States